CLINICAL TRIAL: NCT06091605
Title: Evaluation of Omega Roll Envelope Flap for Soft Tissue Augmentation Around Osseointegrated Dental Implants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Saeed Abd El Aziz, Phd Researcher, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FD-ASU1255
Record Dates: First submitted 2023-09-21; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Soft Tissue Augmentation; Dental Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega roll envelope flap (OREF) technique (Experimental): Patients will undergo peri-implant soft tissue augmentation procedures accompanied by the placement of healing abutments at the uncovering of the inserted osseo-integrated implants, 12 weeks after the initial stage of implant placement.
  Omega roll envelope flap (OREF) technique will be done around the placed healing abutment, then suturing will be done.
  Interventions: Procedure: Soft tissue augmentation around dental implants.
- Envelope flap combined with a sub-epithelial connective tissue graft (Active Comparator): Patients will undergo peri-implant soft tissue augmentation procedures accompanied by the placement of healing abutments at the uncovering of the inserted osseo-integrated implants, 12 weeks after the initial stage of implant placement.
  An envelope split thickness flap will be made at the concerned implant site and a connective tissue graft will be harvested from the tuberosity and then adapted to the placed healing abutment at the surgical site and suturing will be done.
  Interventions: Procedure: Soft tissue augmentation around dental implants.

INTERVENTIONS:
Procedure: Soft tissue augmentation around dental implants. — Soft tissue augmentation around dental implants using Omega roll envelope flap (OREF) technique.
  Other Names: Soft tissue augmentation around dental implants using Envelope flap combined with a sub-epithelial connective tissue graft.

SUMMARY:
Abstract Statement of the problem: Peri-implant soft-tissue augmentation procedures can be broadly divided into two groups, depending on their primary therapeutic objective: (1) Peri-implant soft-tissue phenotype modification and (2) Treatment of peri-implant marginal mucosa defects (PMMDs), also known as peri-implant soft-tissue dehiscences.

Aim of the study: The aim of this study will be to evaluate the efficacy of the Omega roll envelope flap (OREF) technique compared to the conventional envelope split-thickness flap technique combined with an autogenous connective tissue graft, in enhancing Peri-implant soft tissue phenotype defined by the gingival thickness, keratinized tissue width, mucosal margin level and interproximal papilla height around implant.

DETAILED DESCRIPTION:
Materials and Methods: 24 patients complaining of a single missing tooth in the with adjacent intact natural teeth and demanding replacing it with the best possible esthetics will be enrolled and recruited from the outpatient clinic, Faculty of Dentistry, Ain Shams University according to eligibility criteria. They will be randomly allocated to two equal groups. Group A (test group, n=12) will have a single implant placed after receiving non-surgical periodontal therapy and then after 12 weeks at the uncovering of the implant and placement of healing abutment, an Omega roll envelope flap (OREF) technique will be carried out for soft tissue augmentation, while Group B (control group, n=12) same procedures will be done but, soft tissue augmentation will be done by an envelope split-thickness flap combined with a sub-epithelial connective tissue graft. After 3 and 6 months Peri-implant soft tissue phenotype defined by gingival thickness, keratinized tissue width, mucosal margin level and interproximal papilla height around implant will be clinically assessed (1ry outcome). The 2ry outcomes will include comparing between the probing depth and clinical attachment level. Postoperative pain and swelling will be recorded by the patient for the 1st two weeks post-surgically. Postoperative instructions and medication will be given to the patient. All readings will be carried out by a calibrated outcome assessor who will be blinded. Data collected will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Systemically free patients (American Society of Anesthesiologists (ASA) I. Patients between 18 - 50 years of both genders and able to understand the nature of the proposed surgery and to sign the informed consent. Ability to comply with the study related procedures such as maintaining good oral hygiene and attending all follow-up scheduled appointments. Patients who complained of a single missing tooth bounded with two adjacent natural sound teeth diagnosed with clinical periodontal health. Necessity for soft tissue augmentation in a single tooth gap determined by a concavity that was present in the edentulous area or tissues with thin biotype being ≤2 mm or with inadequate width of ≤4mm. Adequate bone width for implant placement without need for bone augmentation (confirmed by a single pre-operative cone-beam computed tomography) (CBCT).

Exclusion Criteria:

* Previous soft tissue augmentation in the area. Need for major soft or hard tissue augmentation procedures. Smokers. Patients taking medications that might affect the healing of soft and hard peri-implant tissues.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Peri-implant soft tissue phenotype | Baseline, 3 Months & 6 Months
  Measured in millimeters, using UNC-15 Periodontal Probe/Endodontic File with rubber stopper,

SECONDARY OUTCOMES:
Postoperative pain | At the day of the procedure and for 14 days (registered before bedtime at a specific time point for each patient)
  Numerical rating scale (Visual analog scale) Scores (0-10)
Postoperative swelling | At the day of procedure and for 7 days (registered before bedtime at specific time point for each patient)
  Numerical rating scale (Visual analog scale) Scores (0-10)
Implant soft tissue deficiency Esthetic Score (IDES) | At 6 months
  Scores of:
  * Soft Tissue Margin (STM) (0-5): 0= No improvement of the PSTD and 5=Complete coverage of the metallic components with the mucosal margin at the same level of the homologous tooth.
  * Peri-implant papillae height (PPH) (0-3): 0=Both papillae are more apical than the healthiest papilla tip of the homologous tooth and 3=Both papillae are at the same level (or more coronal) of the healthiest papilla tip of the homologous tooth.
  * Peri-implant Mucosa (PMC) (0-1): 0=Distinguishable from the adjacent soft tissue and 1=Not distinguishable from the adjacent soft tissue.
  * Peri-implant Mucosa Appearance (PMA) (0-1): 0=Presence of at least one of these conditions: scar tissue, MGJ not-aligned, tissue volume too thin or too thick compared to the adjacent soft tissue or tissue texture not similar to the adjacent soft tissue and 1=Absence of scar tissue, MGJ well aligned, tissue volume in line with the adjacent soft tissue or tissue texture similar to the adjacent soft tissue.
Esthetic satisfaction | At 3 and 6 months
  Numerical rating scale (Visual analog scale) Scores (0-10)
Probing depth | Baseline, 3 Months & 6 Months
  Using UNC-15 Periodontal Probe
Clinical Attachment Level (CAL) | Baseline, 3 Months & 6 Months
  Using UNC-15 Periodontal Probe 0mm= Normal <1-2mm= Stage 1 Periodontitis <3-4mm= Stage 2 Periodontitis >5mm= Stage 3 and 4 Perodontitis

IPD SHARING:
Plan to Share IPD: Undecided